CLINICAL TRIAL: NCT04775862
Title: A Prospective Phase II Study Utilizing Circulating Cell Free DNA (cfDNA) Use in the Detection of RAS Mutations in Patients With Advanced Colorectal Cancer.
Brief Title: A Prospective Study Utilizing Circulating Cell Free DNA (cfDNA) Use in the Detection of RAS Mutations in Patients With Advanced Colorectal Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Guard Health Affairs (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC20/170/R
Record Dates: First submitted 2021-02-21; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Colon Cancer
Keywords: colon cancer; Circulating cell free DNA; Colorectal cancer; NGS
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RAS wild type; investigator choice re-challenge with anti EGFR Rx (Experimental)
  Interventions: Drug: investigator choice re-challenge with anti EGFR Rx
- RAS mutant; investigator choice of SOC third line Rx (Active Comparator)
  Interventions: Drug: investigator choice re-challenge with anti EGFR Rx

INTERVENTIONS:
Drug: investigator choice re-challenge with anti EGFR Rx — Upon second progression, patients will be enrolled into the study as per inclusion criteria and consent, and a cfDNA blood test will be drawn, and RAS status will be examined. If RAS is wildtype, then the investigator will decide whether to re-challenge with an anti EGFR antibody , or give SOC third line chemotherapy (Regorafenib or TAS-102).

SUMMARY:
Colorectal cancer remains the commonest cancer among men, and third commonest among women in Saudi Arabia . Presentation with metastatic disease occurs in almost one third of patients , with 5-year survival decreasing significantly from 90% in stage 1 to 14% once the disease is metastatic . There is enthusiasm in the potential for liquid biopsies to provide easily accessible genetic biomarkers for mutational cancer characterization . Epidermal growth factor receptor (EGFR) monoclonal antibodies are widely used in the treatment of advanced colorectal cancer that do not harbor RAS mutations (RAS wild type). Hence genotyping of oncogenic RAS mutations is essential prior to the initiation of systemic therapy for such patients as the presence of these mutations predict resistance to EGFR targeted antibodies such as Cetuximab and Panitumumab . Detection of such mutations has been done on tissue biopsies with the disadvantage of this being an invasive procedure, and data suggesting that such testing may not be reflective of the true mutational burden of the disease since a single fragment of tissue may be inadequate to reflect the intratumoral heterogeneity. There is increasing evidence suggesting that liquid biopsies or blood based mutational profiling can provide a more comprehensive molecular profile of the disease, and carries the advantage of being minimally invasive. Serial liquid biopsies can act as a tool to identify spatial and temporal heterogeneity predicting response or resistance to targeted agents, and can shed light into the emergence (or disappearance) of specific mutations that may potentially be targeted with newer anti cancer agents .

Circulating cell free DNA (cfDNA) consists of small nucleic acid fragments liberated from cells by rupture, necrosis or apoptosis, and is now increasingly being used to detect RAS (and other) mutations in patients with advanced colorectal cancers. KRAS has remained an "undruggable" target for decades until the most recent evidence that showed a new anticancer drug that targets KRAS G12C mutation.

The investigators aim to perform cfDNA testing on patients with advanced colorectal cancers who have no RAS mutations (and hence start on EGFR inhibitors) as baseline, compare the results with mutational analysis on fresh tumor tissue, and perform cfDNA at first progression to determine what mutations have emerged, and specifically look for KRAS G12C mutation, which can be targeted with a new novel anti cancer drug . These patients will be collected over a 12 month period (with the aim of performing this on at least 100 patients), and followed from diagnosis (with baseline cfDNA) and until progression on EGFR inhibitors (where another cfDNA sample will be taken). A detailed proposal delineating this process will follow once accepted.

This project is unique as it examines mechanisms of resistance to anti-EGFR inhibitors in our patients with advanced colorectal cancers, determines the prevalence of a specific mutation using liquid biopsies and examining cfDNA use, and may have therapeutic implications in facilitating obtaining KRAS G12C inhibitors for such patients.

DETAILED DESCRIPTION:
Colorectal cancer remains the commonest cancer among men, and third commonest among women in Saudi Arabia . Presentation with metastatic disease occurs in almost one third of patients , with 5-year survival decreasing significantly from 90% in stage 1 to 14% once the disease is metastatic . There is enthusiasm in the potential for liquid biopsies to provide easily accessible genetic biomarkers for mutational cancer characterization . Epidermal growth factor receptor (EGFR) monoclonal antibodies are widely used in the treatment of advanced colorectal cancer that do not harbor RAS mutations (RAS wild type). Hence genotyping of oncogenic RAS mutations is essential to be done prior to initiation of systemic therapy for such patients as the presence of these mutations predict resistance to EGFR targeted antibodies such as cetuximab and panitumumab . Treatment of metastatic CRC has become more complex and precision medicine approaches have evolved in recent years with the discovery of new oncogenic (potentially targetable) pathways . The prognosis of metastatic colorectal cancer has improved from 6 months with best supportive care to more than 2 years with multi-agent chemo and targeted therapy including anti EGFR antibodies . Targeting other singling pathways in CRC such as adding vascular endothelial growth factor inhibitors has benefitted patients as well . It is estimated that 55% of patients with metastatic colorectal cancer (mCRC) will have oncogenic mutations in KRAS and NRAS. Detection of such mutations has been done on tissue biopsies with the disadvantage of this being an invasive procedure, and data suggesting that such testing may not be reflective of the true mutational burden of the disease since a single fragment of tissue may be inadequate to reflect the intratumoral heterogeneity. There is increasing evidence suggesting that liquid biopsies or blood based mutational profiling can provide a more comprehensive molecular profile of the disease, and carries the advantage of being minimally invasive. Serial liquid biopsies can act as a tool to identify spatial and temporal heterogeneity predicting response or resistance to targeted agents, and can shed light into the emergence (or disappearance) of specific mutations that may potentially be targeted with newer anti cancer agents . To account for this molecular heterogeneity, the genomic profiles of metastatic colorectal cancer patients should be examined at different time points during the course of therapy using liquid biopsy .

There have been small studies that examined mechanisms of resistance to anti EGFR monoclonal antibodies in mCRC using liquid biopsy. A study of 37 mCRC patients who were treated with cetuximab found that 40% of them developed RAS mutations at progression 10). Another study with limited number of participants examined patients with mCRC treated with panitumumab and found that 9 out of 24 patients (38%) developed KRAS mutations on treatment as a mechanism of acquired resistance to anti EGFR therapy . Furthermore, fewer studies with limited number of patients used liquid biopsy as a biomarker when re-challenging mCRC patients with EGFR monoclonal antibodies. The majority of these studies were retrospective. However, one was the first prospective trial and had a similar protocol to our study. It included 28 patients and reported that 52% of these patients were RAS wildtype at re-challenge with cetuximab - when these patients were exposed to, and progressed on cetuximab in the first line setting. This study showed that re-challenge with cetuximab significantly improved progression free survival when RAS was found to be wild type on circulating tumor DNA(12). One of the limitations of this study was that a single liquid biopsy sample was done (prior to re-challenge with cetuximab) and hence does not display the predicted "switch" of the RAS target, which the investigators plan to study in our trial. Furthermore, a more recent study protocol has been published at BMC Cancer where the investigators plan to study 120 patients and perform liquid biopsy analysis every 3 months while patients are on first line cetuximab. This is to study the evolution of the RAS target, and to correlate this with disease response, as well as help guide therapy with EGFR inhibitors in mCRC patients. However, based on limited data, current guidelines have not yet adopted testing using liquid biopsy and using this strategy to decide on re challenge of anti EGFR therapy in 3rd line setting or not, which is the question investigators would like to answer in this study.

Circulating cell free DNA (cfDNA) consists of small nucleic acid fragments liberated from cells by rupture, necrosis or apoptosis originating from normal and deceased cells, and is now increasingly being used to detect RAS (and other) mutations in patients with advanced colorectal cancers. There is new evidence that G12C RAS mutation can be targeted with a novel anti cancer agent .

the investigators aim to perform cfDNA testing on patients with advanced colorectal cancers who have no RAS mutations i.e wild type (and hence start on EGFR inhibitors - which is standard of care treatment) pre third line therapy. This will help the treating physician decide whether to give these patients with RAS wt status an anti-EGFR monoclonal antibody or standard third line therapy (Regorafenib or TAS-102). These patients will be collected over an 18 month period. The cfDNA test at second progression (i.e prior to third line systemic therapy) will determine whether the subset of patients who may have developed RAS mutation(s) after progression to first line therapy (or other mutations as a mechanism of resistance) with anti - EGFR monoclonal antibodies have switched their RAS status and became wild type. This will support the re-challenge of EGFR inhibitors in the third line setting, and has the potential of changing the colorectal cancer treatment guidelines. Upon this, the principle investigator will decide whether to re-challenge with anti EGFR inhibitor. The investigators aim to study 60 patients in total and have 30 patients at least in the rechallenge (with anti EGFR mAb) group.

Materials and Methods

Patients will have their standard of care (SOC) biopsy of tumor/ metastatic site to confirm diagnosis, and determine RAS status. Once RAS wild type, and primary disease is left sided, these patients will receive standard chemotherapy (choices of FOLFOX, FLOFIRI, CapeOX, XELIRI) with an anti EGFR mAb (cetuximab or panitumumab). Upon progression of disease, second line systemic chemotherapy +/- anti VEGF antibody will be given as per SOC. Upon second progression, patients will be enrolled into the study as per inclusion criteria and consent, and a cfDNA blood test will be drawn, and RAS status will be examined. If RAS is wildtype, then the investigator will decide whether to re-challenge with an anti EGFR antibody (see study schema - figure 1), or give SOC third line chemotherapy (Regorafenib or TAS-102).

Disease assessments will be done every 8 - 12 weeks as per SOC using CT scans, and/or MRI, and will be reported as per RECIST criteria v1.1.

Methods for cfDNA Next Generation Sequencing (NGS) from CRC patients cfDNA extraction Blood samples will be collected in K2EDTA tubes (BD Vacutainer® Blood Collection Tubes, Becton Dickinson, Franklin Lakes, USA) and sent to the Translational Pathology Laboratory. The plasma fraction will be separated from the blood cells by two consecutive rounds of centrifugation for 30 min at room temperature at 1600 × g. The collected plasma was aliquoted and stored at -80 °C until use. cfDNA is extracted from plasma volumes ranging from 0.4 to 5.5 ml using the MagMax Cell-Free Total Nucleic Acid Isolation Kit (Thermo Fisher Scientific, Waltham, USA) according to the manufacturers' instructions. The cfDNA quantity was assessed with the dsDNA HS assay kit by the Qubit 2.0 Fluorometer (Thermo Fisher Scientific). cfDNA quality was assessed with the Agilent Tap Station System (Agilent Technologies, Santa Clara, USA). Only cfDNA samples with a clear fragment size peak between 140-200 bp will be considered for analysis.

NGS library preparation NGS libraries will prepared from 10 ng of cfDNA following the Oncomine™ Pan-Cancer Cell-Free Assay (Thermo Fisher Scientific). Our general library preparation protocol is based on a two-cycle multiplex touch-down PCR reaction with a temperature range from 64 °C to 58 °C, which allowed to amplify target regions and introduce unique molecular identifiers. The resulting tagged amplicons of around 100-140 bp length are then cleaned up using Agencourt AMPure XP (Beckman Coulter, Brea, USA) at a bead to sample ratio of 1.5× and purified products are eluted in 24 μl low TE buffer. A second round of PCR (18 cycles) will be performed in a total volume of 50 μl to amplify the purified amplicons and introduce Ion Torrent™ Tag-Sequencing adapters containing sample-specific barcodes. The resulting library of target DNA fragments will be purified by performing a two-step cleanup using Agencourt AMPure XP (Beckman Coulter) at a bead to sample ratio of 1.15× and 1.0×, respectively. The purified libraries re then diluted 1:1000 and quantified by qPCR using the Ion Universal Quantitation Kit (Thermo Fisher Scientific). The quantified stock libraries are then diluted to 100 pM for downstream template preparation.

Sequencing NGS libraries will be sequenced on an Ion S5™ instrument (Thermo Fisher Scientific) using semiconductor sequencing technology. Briefly, sequencing runs are planned on the Torrent Suite Software™ v5.10, libraries are pooled and loaded on an Ion 540™ chip using the Ion Chef™ instrument (Thermo Fisher Scientific). The loaded chip is then sequenced using 500 flows. Raw data are processed automatically on the Torrent Server™ and aligned to the reference hg19 genome. QC will be performed manually for each sample based on the following metrics; number of reads per sample>15,000,000 (for Oncomine™ Pan-Cancer Cell-Free Assay libraries aries), on-target reads >90%, read uniformity >90%, median molecular coverage >500×, median read coverage >15,000. Tissue NGS libraries are then sequenced according to the manufacturer's instructions. The sequencing data of the QC passing samples are then uploaded in BAM format to the Ion Reporter™ Analysis Server for variant calling and annotation.

Data Analysis For plasma samples variant calling is performed on Ion Reporter™ (IR) Analysis Software v5.10 using the Oncomine™ TagSeq Pan-Cancer Liquid Biopsy w2.0 workflows. The analysis pipeline also includ signal processing, base calling, quality score assignment, adapter trimming, PCR duplicate removal, and control of mapping quality. Coverage metrics for each amplicon is obtained by running the Coverage Analysis Plugin software v5.6 (Thermo Fisher Scientific). Identified variants are only considered if the variant had a molecular coverage of at least three, indicating that the variant is detected in three independent template molecules. Finally, all candidate mutations are manually reviewed using the Integrative Genomics Viewer. Further annotation will be performed by Qiagen QCI platform and in-house oLIMS system.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged >18 years who are diagnosed histologically with advanced/ metastatic colorectal adenocarcinoma.

  * Primary disease must be in left side of colon.
  * ECOG performance status of </= 2.
  * The primary treating physician believes that the patient has a life expectancy of more than 3 months at enrollment.
  * Tumor characteristics at baseline must be RAS/ BRAF wildtype.
  * Must have RECIST measurable disease.
  * Metastatic burden </= 3 organ involvement.
  * Adequate bone marrow, liver and renal function assessed within 14 days before starting systemic treatment.
  * Signed informed consent before any study specific procedures.

Exclusion Criteria:

* Patients with peritoneal metastases.

  * Life expectancy of less than 3 months in the opinion of the investigator.
  * Refusal to consent.
  * Past or current history of malignancy other than colorectal carcinoma, except for curatively treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix.
  * Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-02-21 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Objective response rates (ORR) | 3.5 years
  ORR is defined as the percentage of patients, relative to the total of enrolled subjects, achieving a complete response (CR) or partial response (PR) according to RECIST v1.1 criteria.
Progression-free survival (PFS) | 3.5 years
  PFS is defined as the time from the start of therapy until the first documentation of objective disease progression or death due to any cause, whichever comes first.

SECONDARY OUTCOMES:
Determine proportion of patients with mCRC who are RAS wt after 2nd progression using cfDNA | 3.5 years
Determine the prevalence of RAS G12C mutation via using cfDNA | 3.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ministry of National Guard - Health Affairs, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided